CLINICAL TRIAL: NCT03216278
Title: A Two Part Bioequivalence Study to Compare Two Fixed Dose Combination (FDC) Tablets of Dapagliflozin/Metformin XR 5/500 mg (Part 1) and 10/1000 mg (Part 2) Manufactured at Two Different Plants (Humacao, Puerto Rico and Mount Vernon, US) in Healthy Subjects Under Fasting and Fed Conditions
Brief Title: The Purpose of the Study is to Compare Two Fixed Dose Combination Tablets of Dapagliflozin/Metformin XR in Healthy Subjects Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1691C00016
Record Dates: First submitted 2017-04-07; First posted 2017-07-13 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Healthy Subjects in Fasted and Fed State
Keywords: healthy,; fasted,; fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Treatment A (Experimental): Dapagliflozin/metformin XR 5/500 Mount Vernon Test Product Fed
  Interventions: Drug: Dapagliflozin/metformin XR 5/500mg
- Treatment B (Active Comparator): Dapagliflozin/metformin XR 5/500 Humacao Reference Product Fed
  Interventions: Drug: Dapagliflozin/metformin XR 5/500 mg
- Treatment C (Experimental): Dapagliflozin/metformin XR 5/500 Mount Vernon Test Product Fasted
  Interventions: Drug: Dapagliflozin/metformin XR 5/500mg
- Treatment D (Active Comparator): Dapagliflozin/metformin XR 5/500 Humacao Reference Product Fasted
  Interventions: Drug: Dapagliflozin/metformin XR 5/500mg
- Treatment E (Experimental): Dapagliflozin/metformin XR 10/1000 Mount Vernon Test Product Fed
  Interventions: Drug: Dapagliflozin/metformin XR 10/1000mg
- Treatment F (Active Comparator): Dapagliflozin/metformin XR 10/1000 Humacao Reference Product Fed
  Interventions: Drug: Dapagliflozin/metformin XR 10/1000mg
- Treatment G (Experimental): Dapagliflozin/metformin XR 10/1000 Mount Vernon Test Product Fasted
  Interventions: Drug: Dapagliflozin/metformin XR 10/1000mg
- Treatment H (Active Comparator): Dapagliflozin/metformin XR 10/1000 Humacao Reference Product Fasted
  Interventions: Drug: Dapagliflozin/metformin XR 10/1000mg

INTERVENTIONS:
Drug: Dapagliflozin/metformin XR 5/500mg — Tablets for oral administration, once daily, once per treatment period
  Other Names: Mt Vernon plant
  Arms: Treatment A
Drug: Dapagliflozin/metformin XR 5/500 mg — Tablets for oral administration, once daily, once per treatment period
  Other Names: Humacao plant
  Arms: Treatment B
Drug: Dapagliflozin/metformin XR 5/500mg — Tablets for oral administration, once daily, once per treatment period
  Other Names: Dapagliflozin/metformin XR 5/500mg Mount Vernon plant
  Arms: Treatment C
Drug: Dapagliflozin/metformin XR 5/500mg — Tablets for oral administration, once daily, once per treatment period
  Other Names: Humacao plant
  Arms: Treatment D
Drug: Dapagliflozin/metformin XR 10/1000mg — Tablets for oral administration, once daily, once per treatment period
  Other Names: Mount Vernon plant
  Arms: Treatment E
Drug: Dapagliflozin/metformin XR 10/1000mg — Tablets for oral administration, once daily, once per treatment period
  Other Names: Humacao plant
  Arms: Treatment F
Drug: Dapagliflozin/metformin XR 10/1000mg — Tablets for oral administration, once daily, once per treatment period
  Other Names: Dapagliflozin/metformin XR 10/1000mg Mount Vernon plant
  Arms: Treatment G
Drug: Dapagliflozin/metformin XR 10/1000mg — Tablets for oral administration, once daily, once per treatment period
  Other Names: Dapagliflozin/metformin XR 10/1000mg Humacao plant
  Arms: Treatment H

SUMMARY:
This is a bioequivalence study of two doses of the dapagliflozin/metformin XR tablet manufactured at two different plants.

DETAILED DESCRIPTION:
This is a two part, open-label, randomized, 4-period, 4-treatment (per study part) crossover study in healthy subjects (males and females of non-childbearing potential), performed at a single study center, conducted to establish the bioequivalence of 2 strengths of dapagliflozin/metformin XR tablets manufactured at two different plants.

ELIGIBILITY:
Inclusion criteria

1. Provision of signed and dated, written informed consent prior to any study-specific procedures
2. Healthy male and female subjects aged 18 - 50 years with suitable veins for cannulation or repeated venipuncture
3. Females must have a negative serum pregnancy test at screening and negative urine pregnancy test on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling 1 of the following criteria:

   * Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post menopausal range
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation
4. Have a body mass index (BMI) between 18.50 and 24.90 kg/m2 inclusive [15% variance on the upper limit is permitted (i.e., up to 28.63 kg/m2)] and weigh between 50 and 100 kg inclusive at screening

Exclusion Criteria

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the investigator
5. Any clinically significant abnormal findings in vital signs, as judged by the investigator
6. Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) as judged by the investigator
7. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) antibody
8. Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
9. Total bilirubin >2.0 mg/dL (34.2 µmol/L)
10. Known or suspected history of drug abuse, as judged by the investigator
11. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose.

    Note: Subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
12. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening
13. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to dapagliflozin/metformin XR.
14. Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
15. Positive screen for drugs of abuse or alcohol at screening or on each admission to the study center
16. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP
17. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, vitamins and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life Note: Hormonal replacement therapy is allowed for females.
18. Known or suspected history of alcohol abuse or excessive intake of alcohol, as judged by the investigator
19. Inclusion of any AstraZeneca or study site employee or their close relatives
20. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements
21. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Part 1 - Area under the plasma concentration versus time curve (AUC) for each analyte and each state | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  To demonstrate the bioequivalence of dapagliflozin/metformin XR 5/500 mg manufactured at Mount Vernon plant and dapagliflozin/metformin XR 5/500 mg manufactured at Humacao plant in metformin and in dapagliflozin plasma concentrations for the fed state and, separately, the fasted state.
Part 2 - Area under the plasma concentration versus time curve (AUC) for each analyte and each state | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  To demonstrate the bioequivalence of dapagliflozin/metformin XR 10/1000 mg manufactured at Mount Vernon plant and dapagliflozin/metformin XR 10/1000 mg manufactured at Humacao plant in metformin and dapagliflozin plasma concentrations for the fed state and, separately, the fasted state.
Part 1 - Peak Plasma Concentration (Cmax) for each analyte and each state | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  To demonstrate the bioequivalence of dapagliflozin/metformin XR 5/500 mg manufactured at Mount Vernon plant and dapagliflozin/metformin XR 5/500 mg manufactured at Humacao plant in metformin and in dapagliflozin plasma concentrations for the fed state and, separately, the fasted state.
Part 2 - Peak Plasma Concentration (Cmax) for each analyte and each state | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  To demonstrate the bioequivalence of dapagliflozin/metformin XR 10/1000 mg manufactured at Mount Vernon plant and dapagliflozin/metformin XR 10/1000 mg manufactured at Humacao plant in metformin and in dapagliflozin plasma concentrations for the fed state and, separately, the fasted state.

SECONDARY OUTCOMES:
Area under plasma concentration - time curve from time zero to infinity (AUC) | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  Measurements of AUC from time zero to infinity for dapagliflozin and metformin when administered as single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants both fed and fasted states.
Adverse events | 10,5 weeks
  To evaluate the safety of single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants both fed and fasted states by assessing the number of subjects with adverse events.
Blood pressure | 10,5 weeks
  To evaluate the safety of single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants both fed and fasted states by assessing changes from baseline in mmHg of systolic and diastolic blood pressure.
Electrocardiogram (ECG) | 10,5 weeks
  To evaluate the safety of single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants both fed and fasted states by assessing changes from baseline in overall ECG evaluation.
Time to reach maximum plasma concentration (tmax) | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  Measurements of tmax for dapagliflozin and metformin when administered in both fed and fasted states as single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  Measurements of half-life associated with terminal slope (t½λz) for dapagliflozin and metformin when administered in both fed and fasted states as single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants.
Terminal elimination rate constant (λz) | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  Measurements of terminal elimination rate constant (λz) for dapagliflozin and metformin when administered in both fed and fasted states as single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants.
Apparent total body clearance after extravascular administration (CL/F) | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  Measurements of apparent total body clearance after extravascular administration (CL/F) for dapagliflozin and metformin when administered in both fed and fasted states as single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | Based on pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose sampling times
  Measurements of apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) for dapagliflozin and metformin when administered in both fed and fasted states as single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants.
Laboratory assessments - hematology | 10,5 weeks
  To evaluate the safety of single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants both fed and fasted states by assessing changes from baseline in hematology.
Heart rate | 10,5 weeks
  To evaluate the safety of single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants both fed and fasted states by assessing changes from baseline in heart rate measured as beats per minute.
Laboratory assessments - clinical chemistry | 10,5 weeks
  To evaluate the safety of single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants both fed and fasted states by assessing changes from baseline in clinical chemistry.
Laboratory assessments - urinalysis | 10,5 weeks
  To evaluate the safety of single doses of dapagliflozin/metformin 5/500 mg or 10/1000 mg formulation from both the Mount Vernon and Humacao plants both fed and fasted states by assessing changes from baseline in urinalysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Aparecida de Goiânia, Brazil

IPD SHARING:
Plan to Share IPD: Yes